CLINICAL TRIAL: NCT02705287
Title: Vitamin D Dynamics in Pregnant Women and Non-Pregnant Women of Reproductive Age
Brief Title: Vitamin D Dynamics in Women
Status: Recruiting | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: IRB # 1509005821; RSRB00057617 (Other: University of Rochester)
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy
Keywords: vitamin D; half life; kinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples and extracted DNA sample (biospecimen retention will be both with and without DNA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Vitamin D dynamics- pregnant: Pregnant women recruited to measure Vitamin D dynamics during pregnancy.
  Interventions: Other: Vitamin D dynamics-pregnant
- Vitamin D dynamics-nonpregnant: Non-pregnant women recruited to measure Vitamin D dynamics.
  Interventions: Other: Vitamin D dynamics-nonpregnant

INTERVENTIONS:
Other: Vitamin D dynamics-pregnant — tracer dose of deuterated vitamin D3
  Groups: Vitamin D dynamics- pregnant
Other: Vitamin D dynamics-nonpregnant — tracer dose of deuterated vitamin D3
  Groups: Vitamin D dynamics-nonpregnant

SUMMARY:
The goal of this project is to utilize stable isotopically labeled vitamin D3 and state of the art mass spectrometric methodology to assess vitamin D dynamics during pregnancy in relation to relation to obesity and vitamin D binding protein genotype. At the conclusion of this study, the investigators will have obtained novel information on the absorption and utilization of vitamin D in women and the degree to which vitamin D utilization during pregnancy is impacted by genetic ancestry, vitamin D binding protein concentration and genotype and by excess adiposity. The long-term goal is to better understand the unique metabolism of vitamin D during pregnancy.

DETAILED DESCRIPTION:
Nearly 30% of US women are either vitamin D insufficient or deficient. Vitamin D inadequacy during gestation is increasingly linked to adverse birth outcomes including preterm birth, the risk of cesarean section and placental and pregnancy-associated infections. At this time the Institute of Medicine (IOM) has not advocated any increase in vitamin D intake across gestation but this remains controversial in large part due to insufficient information on the basic physiology of vitamin D. Pregnancy induces dramatic changes in regulation of vitamin D. The investigators hypothesize that increased maternal, placental, and fetal vitamin D requirements during late gestation will result in an increase in vitamin D absorption and a decrease in the half-life of both vitamin D3 and 25-hydroxyvitamin D. The fetus is entirely dependent on maternal vitamin D to meet its requirements for this nutrient. Maternal vitamin D is thought to be passively transferred across the placenta to the fetus given that neonatal concentrations of 25(OH)D are at least 20-30% lower than maternal 25(OH)D concentrations. To date, much of what is known about vitamin D absorption and utilization in humans has been extrapolated from early radiotracer studies in adult men and non-pregnant women and there are no in vivo data to determine if maternal vitamin D3 or maternal 25(OH)D3, or both, can be transferred across the placenta to the fetus

The specific aims of this project are to:

1. To characterize the impact of pregnancy on the absorption of vitamin D3, conversion into 25(OH)D3, and serum half-life of 25OH)D3 in pregnant and non-pregnant women using tri-deuterated vitamin D3, state of the art UHPLC-MS/MS methodology and mathematical modeling.
2. To study the impact of obesity on vitamin D kinetics and the D content of serum and adipose tissue in pregnant and non-pregnant women.
3. To evaluate the impact of genetic ancestry on vitamin D kinetics and the D content of serum and adipose tissue in pregnant and non-pregnant women.

ELIGIBILITY:
Inclusion Criteria (Non-pregnant and pregnant participants participants):

* Self-reported White and Black women
* Age 20-39
* Body mass index (BMI) 1or pre-pregnancy BMI (If currently pregnant) either 18.5-24.9 kg/m2 or greater than or equal to 30 kg/m2

Inclusion Criteria (Additional criteria for pregnant participants):

* Singleton pregnancy
* Recruited in first trimester, second trimester, or third trimester
* No pregnancy complications

Exclusion Criteria (Non-pregnant and pregnant participants):

* BMI or pre-pregnancy BMI <18.5 kg/m2
* Human immunodeficiency virus (HIV) infection
* Diagnosed eating disorder
* Malabsorption disease
* Diabetes
* Elevated diastolic blood pressure (>110 mm/Hg)
* Steroid use
* Substance abuse history
* Current use of medications known to influence vitamin D or calcium homeostasis
* Plans to travel to lower latitude during the 20-day study period
* Plans to become pregnant during the study period (non-pregnant only)
* Refuses to discontinue tanning bed use during study period
* Refuses to discontinue vitamin or mineral supplement use during study period (non-pregnant only)

Exclusion Criteria (Additional criteria for pregnant participants):

* Gestational diabetes
* Pregnancy hypertension

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women and non-pregnant women of reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Impact of pregnancy on serum vitamin D absorption | Across 40 days study period
  A baseline blood sample (20 mL) will be obtained for analysis of the baseline concentrations of indicators of vitamin D status. Each woman will be asked to ingest two pieces of toast onto which a dose of 35 μg of [6,19,19-d3]-vitamin D3 has been added. Women will return to the at 4 hour, 8 hour, Day 2, 10, 25, and 40 (± 2 days) for an additional blood sample (15 mL each) to assess the disappearance of the tri-deuterated D3, conversion into 25(OH)D3, and serum half-life of 25(OH)D3.
Impact of obesity on vitamin D absorption | Across 40 days study period
  A baseline blood sample (20 mL) will be obtained for analysis of the baseline concentrations of indicators of vitamin D status. Each woman will be asked to ingest two pieces of toast onto which a dose of 35 μg of [6,19,19-d3]-vitamin D3 has been added. Women will return to the at 4 hour, 8 hour, Day 2, 10, 25, and 40 (± 2 days) for an additional blood sample (15 mL each) to assess the disappearance of the tri-deuterated D3, conversion into 25(OH)D3, and serum half-life of 25(OH)D3. Body composition measure using Bioelectrical Impedance Analysis (BIA) will be conducted on Day 0 for all participants and Day 40 for he pregnant participants to obtain information on BMI and fat mass. Adipose tissue (<1 gram) will be extracted using needle biopsy from the upper buttock area on all participants for D content analysis.
Impact of ancestry on serum vitamin D absorption | Across 40 days study period
  A baseline blood sample (20 mL) will be obtained for analysis of the baseline concentrations of calcitropic hormones and indicators of vitamin D status. Each woman will be asked to ingest one quarter piece of toast onto which a dose of 35 ug of [6,19,19-d3]-vitamin D3 has been added. Women will return to the at 4 hour, 8 hour, Day 1, 3, 10, 25, and 40 (± 2 days) for an additional blood sample (15 mL each) to assess the disappearance of the tri-deuterated D3, conversion into 25(OH)D3, and serum half-life of 25(OH)D3. DNA will be extracted to perform ancestry genotyping and determine vitamin D binding protein genotypes.

SECONDARY OUTCOMES:
Placental protein quantification | Across 40 days study period
  At delivery placental tissue will be collected for evaluation of placental mRNA expression and protein abundance of CYP2R1, CYP24A1 and CYP27B1 following methods we, and others have published. This will help us obtain data on placental contributions to D utilization to inform our mathematical model and hypotheses.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O. O'Brien, PhD, Principal Investigator — Cornell University; Eva Pressman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, 518 Hylan Building, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No